CLINICAL TRIAL: NCT04894175
Title: Association Between Treatment Perception and Treatment Adherence in Obstructive Sleep Apnea Patients Treated by Continuous Positive Airway Pressure (SEMSAS Study)
Brief Title: Association Between Treatment Adherence and Treatment Adherence in Sleep Apnea (SEMSAS)
Acronym: SEMSAS
Status: Completed | Type: Observational
Sponsor: Thibaut Gentina (Industry)
Responsible Party: Sponsor-Investigator, Thibaut Gentina, Principal investigator, Auxilair
Organization: Auxilair (Industry)
Other Study IDs: 20.09.01.60526
Record Dates: First submitted 2021-05-12; First posted 2021-05-20 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of the study is to define an optimal threshold of the SEMSA-15 scale for obstructive sleep apnea (OSA) perception in patients with OSA to predict 3-month and 1-year continuous positive airway pressure adherence.

ELIGIBILITY:
Inclusion Criteria:

* Obstructive Sleep apnea diagnosed, whatever the initial severity and treated with CPAP
* Voluntary patient
* patient in the national healthcare insurance system

Exclusion Criteria:

* Patient with central sleep apnea
* Treatment other than CPAP
* Person with liberty privation or under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population will be screened by clinicians (pulmonologists) in ambulatory medicine
Sampling Method: Non-Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Continuous positive airway pressure adherence | 3-month
  To define an optimal threshold for the Self-efficacy Measure for Sleep Apnea (SEMSA-15) scale to predict 3-month CPAP adherence
Continuous positive airway pressure adherence | 1-year
  To define an optimal threshold for the Self-efficacy Measure for Sleep Apnea (SEMSA-15) scale to predict 1-year CPAP adherence

SECONDARY OUTCOMES:
To compute an overall score to predict CPAP adherence | 3-month and 1-year
  Use Self-efficacy Measure for Sleep Apnea (SEMSA-15) scale and socio-economics parameter from patients to improve CPAP adherence prediction
To study the impact of health litteracy on CPAP adherence | 3-month and 1-year
  Use of Health Litteracy Questionnaire HLQ
To study the impact of precariousness on CPAP adherence | 3-month and 1-year
  Use of Deprivation in Primary Care (DIPCARE-Q) questionnaire
To study the impact of patient quality of life on CPAP adherence | 3-month and 1-year
  Use of simplified Short-Form (SF-36) questionnaire for quality of life (SF-12 questionnaire)
To construct an overall predictive model of CPAP adherence | 3-month and 1-year
  CPAP Adherence
To assess the interactions between CPAP adherence trajectories and patients parameters | 3-month and 1-year
  CPAP adherence trajectories
to assess the improvement of quality of life according to health litteracy and precariousness | 1-year
  Quality of life
Define patient phenotype according all collected variables | At inclusion
  Clinical and socio-demographic phenotype at CPAP initiation

CONTACTS AND LOCATIONS:
Overall Officials: Thibaut Gentina, MD, Principal Investigator — Hopital La Louvière
Locations (1):
- Gentina, Lille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gentina T, Micoulaud-Franchi JA, Gentina E, Wang KP, Pepin JL, Bailly S. Association between Self-Efficacy and 1-Year Continuous Positive Airway Pressure Adherence Trajectories: Insight from the SEMSAS Study. Ann Am Thorac Soc. 2025 Dec;22(12):1942-1950. doi: 10.1513/AnnalsATS.202502-231OC. PMID 40680220